CLINICAL TRIAL: NCT01164371
Title: Gender Differences in the Development and Prognosis of Coronary Disease Where Initial Disease Manifestation is Stable Angina, Myocardial Infarction or Unheralded Coronary Death: A CALIBER Study Using Linked GPRD-MINAP Data
Brief Title: Gender Differences in the Development, Treatment and Prognosis of Coronary Disease: A CALIBER Study
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Barts and the London School of Medicine and Dentistry (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Julie George, NIHR Doctoral Fellow, University College, London
Other Study IDs: CALIBER-09-05
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Disease; Cardiovascular Disease
Keywords: coronary disease; cardiovascular disease; cardiovascular risk; cardiovascular risk management; primary care; angina; stable angina; angina pectoris; acute coronary syndrome; coronary death; unheralded acute coronary syndrome; unheralded coronary death; gender differences; sex differences; myocardial infarction; ST elevation myocardial infarction; non ST elevation myocardial infarction; STEMI; nSTEMI; unstable angina
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Angina Pectoris; Angina, Stable; Acute Coronary Syndrome; Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Initial presentation of coronary disease - Stable angina: Patients whose initial symptomatic presentation of coronary disease is stable angina (either diagnosis or symptoms)
- Initial presentation of coronary disease - ACS: Patients whose initial symptomatic presentation of coronary disease is acute coronary syndrome (ST-elevation myocardial infarction [STEMI], non-STEMI [nSTEMI] or unstable angina) without prior stable angina or symptoms of stable angina
- Initial presentation of coronary disease - Coronary death: Patients whose initial symptomatic manifestation of coronary disease is coronary death with no prior diagnosis of stable angina (or symptoms of stable angina) or diagnosis of acute coronary syndrome
- Initial presentation of coronary disease - None: Patients without symptomatic presentation of coronary disease, either alive or dead from non-coronary cause

SUMMARY:
The initial manifestation of symptomatic coronary disease can range from angina (or symptoms of angina), unheralded acute coronary syndrome (ACS), or unheralded coronary death. A better understanding of gender differences in initial presentation of coronary disease and the rate and predictors of progression to subsequent stages in coronary disease could help to identify which gender- specific factors might reduce or slow transition to more serious disease states and improve outcomes. The investigators' research focuses on the role primary care management of cardiovascular risk factors plays in gender differences in the progression to subsequent disease states and to mortality.

DETAILED DESCRIPTION:
The initial manifestation of symptomatic coronary disease can range from angina (or symptoms of angina), unheralded acute coronary syndrome, or unheralded coronary death. Gender differences in initial presentation of coronary disease and the rate and predictors of progression to subsequent stages in coronary disease are not well understood. Furthermore, while the management of coronary risk factors in primary care is hypothesized to play a key role in the rate and timing of such transitions, little is known about the impact such management has on gender differences these transitions and outcomes.

Study Objectives:

1. To determine gender differences in probabilities of transitions from symptom-free state to mortality for each of three patient coronary disease pathways, where the initial disease manifestation is angina, myocardial infarction or unheralded coronary death.
2. To determine the role management of coronary risk factors in primary care has in explaining any gender differences in transitions from symptom-free state to mortality for each of the three patient coronary disease pathways.

A statistical analytic protocol for the first part of this study, comparing patients with unheralded coronary death to patients free of symptomatic coronary disease, dated June 2010, is available on request. A second statistical analytic protocol for the second part of this study, comparing initial presentation of coronary disease, within a framework of competing risks of atherosclerotic disease, dated December 2011, is available on request.

This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

ELIGIBILITY:
Inclusion Criteria:

* as above

Exclusion Criteria:

* patients with a history of ischaemic heart disease, heart failure, cerebrovascular disease, peripheral arterial disease or congenital coronary anomalies, prior to entry into the cohort
* patients with symptoms of chest pain in the 6 months prior to cohort entry
* patients < 35 or >100 years of age after eligibility for entry to the cohort

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all adults aged 35 or over in General Practice Research Database (GPRD), registered with an up-to-standard practice with at least 1 year of continuous follow-up.
  Further details on defining up-to-standard practices within GPRD are available from http://www.gprd.com/home/
Sampling Method: Non-Probability Sample
Enrollment: 1758584 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
coronary mortality (ICD 10 I20-I25) | up to 15 years from entry into cohort
  coronary mortality, following symptom free state, diagnosed angina or acute coronary syndrome

SECONDARY OUTCOMES:
stable angina | up to 15 years from entry into cohort
  diagnosis of angina following symptom free state
acute non-fatal acute coronary syndrome, comprising ST elevation myocardial infarction, non-ST elevation myocardial infarction, and unstable angina | up to 15 years from entry into cohort
  acute coronary syndrome following either symptom-free state (unheralded) or stable angina

CONTACTS AND LOCATIONS:
Overall Officials: Julie George, MSc, Principal Investigator — University College, London

IPD SHARING:
Plan to Share IPD: No
Permissions to used anonymised linked data from data owners prohibit further sharing of the data

REFERENCES:
- [Background] Richards H, McConnachie A, Morrison C, Murray K, Watt G. Social and gender variation in the prevalence, presentation and general practitioner provisional diagnosis of chest pain. J Epidemiol Community Health. 2000 Sep;54(9):714-8. doi: 10.1136/jech.54.9.714. PMID 10942455
- [Background] Hemingway H, Langenberg C, Damant J, Frost C, Pyorala K, Barrett-Connor E. Prevalence of angina in women versus men: a systematic review and meta-analysis of international variations across 31 countries. Circulation. 2008 Mar 25;117(12):1526-36. doi: 10.1161/CIRCULATIONAHA.107.720953. Epub 2008 Mar 17. PMID 18347213
- [Background] Hemingway H, McCallum A, Shipley M, Manderbacka K, Martikainen P, Keskimaki I. Incidence and prognostic implications of stable angina pectoris among women and men. JAMA. 2006 Mar 22;295(12):1404-11. doi: 10.1001/jama.295.12.1404. PMID 16551712
- [Background] Buckley BS, Simpson CR, McLernon DJ, Murphy AW, Hannaford PC. Five year prognosis in patients with angina identified in primary care: incident cohort study. BMJ. 2009 Aug 6;339:b3058. doi: 10.1136/bmj.b3058. PMID 19661139
- [Background] Daly C, Clemens F, Lopez Sendon JL, Tavazzi L, Boersma E, Danchin N, Delahaye F, Gitt A, Julian D, Mulcahy D, Ruzyllo W, Thygesen K, Verheugt F, Fox KM; Euro Heart Survey Investigators. Gender differences in the management and clinical outcome of stable angina. Circulation. 2006 Jan 31;113(4):490-8. doi: 10.1161/CIRCULATIONAHA.105.561647. PMID 16449728
- [Background] Murabito JM, Evans JC, Larson MG, Levy D. Prognosis after the onset of coronary heart disease. An investigation of differences in outcome between the sexes according to initial coronary disease presentation. Circulation. 1993 Dec;88(6):2548-55. doi: 10.1161/01.cir.88.6.2548. PMID 8252666
- [Background] Yawn BP, Wollan PC, Jacobsen SJ, Fryer GE, Roger VL. Identification of women's coronary heart disease and risk factors prior to first myocardial infarction. J Womens Health (Larchmt). 2004 Dec;13(10):1087-100. doi: 10.1089/jwh.2004.13.1087. PMID 15650342
- [Background] Champney KP, Frederick PD, Bueno H, Parashar S, Foody J, Merz CN, Canto JG, Lichtman JH, Vaccarino V; NRMI Investigators. The joint contribution of sex, age and type of myocardial infarction on hospital mortality following acute myocardial infarction. Heart. 2009 Jun;95(11):895-9. doi: 10.1136/hrt.2008.155804. Epub 2009 Jan 15. PMID 19147625
- [Background] Vaccarino V, Parsons L, Peterson ED, Rogers WJ, Kiefe CI, Canto J. Sex differences in mortality after acute myocardial infarction: changes from 1994 to 2006. Arch Intern Med. 2009 Oct 26;169(19):1767-74. doi: 10.1001/archinternmed.2009.332. PMID 19858434
- [Background] MacIntyre K, Stewart S, Capewell S, Chalmers JW, Pell JP, Boyd J, Finlayson A, Redpath A, Gilmour H, McMurray JJ. Gender and survival: a population-based study of 201,114 men and women following a first acute myocardial infarction. J Am Coll Cardiol. 2001 Sep;38(3):729-35. doi: 10.1016/s0735-1097(01)01465-6. PMID 11527625
- [Derived] George J, Rapsomaniki E, Pujades-Rodriguez M, Shah AD, Denaxas S, Herrett E, Smeeth L, Timmis A, Hemingway H. How Does Cardiovascular Disease First Present in Women and Men? Incidence of 12 Cardiovascular Diseases in a Contemporary Cohort of 1,937,360 People. Circulation. 2015 Oct 6;132(14):1320-8. doi: 10.1161/CIRCULATIONAHA.114.013797. Epub 2015 Sep 1. PMID 26330414
- [Derived] Rapsomaniki E, Timmis A, George J, Pujades-Rodriguez M, Shah AD, Denaxas S, White IR, Caulfield MJ, Deanfield JE, Smeeth L, Williams B, Hingorani A, Hemingway H. Blood pressure and incidence of twelve cardiovascular diseases: lifetime risks, healthy life-years lost, and age-specific associations in 1.25 million people. Lancet. 2014 May 31;383(9932):1899-911. doi: 10.1016/S0140-6736(14)60685-1. PMID 24881994
- See also: CArdiovascular disease research Linking Bespoke studies and Electronic Records — http://www.caliberresearch.org